CLINICAL TRIAL: NCT00706277
Title: Effect of Total Intravenous Anesthesia and Balanced Anesthesia on Postoperative Lung Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Arnulf Benzer, TILAK A-6020 Innsbruck, Anichstr. 35 AUSTRIA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-007161-25
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Lung Function
Keywords: forced vital capacity; forced expired volume in 1 s
MeSH Terms: interventions — Propofol; Remifentanil; Fentanyl; Sevoflurane; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TIVA (Active Comparator): patients receiving total intravenous anesthesia (TIVA)
  Interventions: Drug: propofol; Drug: remifentanil
- balanced (Active Comparator): patients receiving balanced anesthesia
  Interventions: Drug: propofol; Drug: fentanyl; Drug: Sevoflurane/Nitrous Oxide

INTERVENTIONS:
Drug: propofol — propofol 2mg/kg for induction of anesthesia; followed by propofol 6 mg/kg/hour
  Arms: TIVA
Drug: propofol — propofol 2mg
  Arms: balanced
Drug: remifentanil — remifentanil 0,25mcg/kg/hour
  Arms: TIVA
Drug: fentanyl — fentanyl 100mcg
  Arms: balanced
Drug: Sevoflurane/Nitrous Oxide — maintenance of anesthesia with sevoflurane and nitrous oxide
  Arms: balanced

SUMMARY:
The aim of the study is to investigate the effects of total intravenous anesthesia (TIVA; propofol, remifentanil) and balanced anesthesia (BAL; induction with propofol and fentanyl; maintenance of anesthesia with sevoflurane and nitrous oxide) on pulmonary function 30 minutes after emergence from the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* BMI normal

Exclusion Criteria:

* lung disease
* Nicotine abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
FEV1 forced expiratory volume; FVC forced vital capacity | preoperative, 30 minutes postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Benzer, MD, Principal Investigator — TILAK Hospitals
Locations (1):
- TILAK Hospitals, Innsbruck, Austria

REFERENCES:
- [Background] Gunnarsson L, Lindberg P, Tokics L, Thorstensson O, Thorne A. Lung function after open versus laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 1995 Apr;39(3):302-6. doi: 10.1111/j.1399-6576.1995.tb04066.x. PMID 7793205
- [Background] Regli A, von Ungern-Sternberg BS, Reber A, Schneider MC. Impact of spinal anaesthesia on peri-operative lung volumes in obese and morbidly obese female patients. Anaesthesia. 2006 Mar;61(3):215-21. doi: 10.1111/j.1365-2044.2005.04441.x. PMID 16480344
- [Background] Natalini G, Franceschetti ME, Pletti C, Recupero D, Lanza G, Bernardini A. Impact of laryngeal mask airway and tracheal tube on pulmonary function during the early postoperative period. Acta Anaesthesiol Scand. 2002 May;46(5):525-8. doi: 10.1034/j.1399-6576.2002.460509.x. PMID 12027846